CLINICAL TRIAL: NCT05465954
Title: Efficacy and Safety Study of Neoadjuvant Efineptakin Alfa (NT-I7) and Pembrolizumab in Recurrent Glioblastoma
Brief Title: Efineptakin Alfa and Pembrolizumab for the Treatment of Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: NeoImmuneTech (Industry); Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210706; NCI-2022-05515 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-011200 (Other: Mayo Clinic Institutional Review Board); R01CA288862 (NIH)
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: High Grade Astrocytic Tumor; Recurrent Glioblastoma, IDH-Wildtype; Recurrent Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Specimen Handling; efineptakin alfa; gosha-jinki-gan; pembrolizumab; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (efineptakin alfa, pembrolizumab) (Experimental): BEFORE SURGERY: Patients receive pembrolizumab IV over 30 minutes and efineptakin alfa IM on day 1. Patients then undergo surgery 1 week later.
  AFTER SURGERY: Patients receive pembrolizumab IV over 30 minutes and efineptakin alfa IM on day 1 of each cycle. Cycles repeat every 42 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Patients undergo MRI or CT at baseline and on study. Patients also undergo tumor biopsy at baseline and blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Biological: Efineptakin alfa; Biological: Pembrolizumab; Procedure: Biopsy

INTERVENTIONS:
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Efineptakin alfa — Given IM
  Other Names: GX-I7; Hyleukin-7 (TM); Il-7 Hybrid Fc; IL-7-hyFc; NT-I7; rhIL-7-hyFc; TJ 107; TJ-107; TJ107
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx

SUMMARY:
This phase II trial tests the safety and side effects of efineptakin alfa and pembrolizumab in treating patients with glioblastoma that has come back (recurrent). Efineptakin alfa is an immunotherapy drug that works by helping the immune system fight tumor cells. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving efineptakin alfa and pembrolizumab may kill more tumor cells in patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of pembrolizumab + efineptakin alfa (NT-I7) in combination with surgery in patients with recurrent glioblastoma multiforme (GBM) using the rate of overall survival at 9 months.

SECONDARY OBJECTIVES:

I. To assess progression-free survival in recurrent GBM patients treated with pembrolizumab + NT-I7 in combination with surgery.

II. To determine the objective response rate in recurrent GBM patients treated with pembrolizumab + NT-I7 in combination with surgery.

III. To assess changes in absolute lymphocyte counts (ALC) over time in recurrent GBM patients treated with pembrolizumab + NT-I7 in combination with surgery.

TERTIARY OBJECTIVES:

I. To assess the adverse event (AE) and toxicity profile of pembrolizumab + NT-I7 in combination with surgery in patients with recurrent GBM.

II. To assess the anti-glioma immune response in patients with recurrent GBM, before and after pembrolizumab and NT-I7 treatment, including assessment of cytokine profiling, immune cell phenotyping, function, and activation in the pre/post-treatment blood and tumor tissue when available.

III. To test tumor mutation burden on tumor/immune cells by validated comprehensive genomic profiling.

IV. To evaluate the changes for tumor microenvironment (TME) post pembrolizumab and NT-I7 and their correlations with treatment response and survival.

V. To evaluate tumor infiltrating lymphocytes (CD4, CD8, Treg, etc) in the tumor tissue pre- and post-treatment (when available).

VI. To assess changes in repertoire breadth and clonality by T-cell receptor (TCR) sequencing.

VII. To explore potential tissue and blood biomarkers that may predict response.

OUTLINE:

BEFORE SURGERY: Patients receive pembrolizumab intravenously (IV) over 30 minutes and efineptakin alfa intramuscularly (IM) on day 1. Patients then undergo surgery 1 week later.

AFTER SURGERY: Patients receive pembrolizumab IV over 30 minutes and efineptakin alfa IM on day 1 of each cycle. Cycles repeat every 42 days for 2 years in the absence of disease progression or unacceptable toxicity.

Patients undergo magnetic resonance imaging (MRI) or computed tomography (CT) at baseline and on study. Patients also undergo tumor biopsy at baseline and blood sample collection on study.

After completion of study treatment, patients are followed up at 30 days and every 2-3 months until disease progression (if applicable), and then every 6 months for up to 5 years from study registration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Disease characteristics:

  * Tissue-confirmed progressive or recurrent World Health Organization (WHO) Grade IV IDH wildtype glioblastoma (including molecular glioblastoma and gliosarcoma)
  * Previously treated with maximum feasible resection or biopsy, radiation, and temozolomide
* Have an enhancing mass on magnetic resonance imaging (MRI) amenable to resection or biopsy of the tumor (as determined by the neurosurgeon pre-operatively) and histological diagnosis of glioblastoma from a prior biopsy or surgery
* Willing to undergo clinically indicated biopsy and/or resection of their glioblastoma at Mayo Clinic in Rochester, Minnesota (MN).
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1 and Karnofsky Performance Scale (KPS) >= 70 NOTE: PS must be assessed (again) within 7 days prior to first dose of study drug
* Hemoglobin >= 9.0 g/dL (obtained =< 15 days prior to registration) (without transfusion or erythropoietin [EPO] dependency =< 7 days prior to assessment)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 15 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 15 days prior to registration)
* Creatinine =< 1.5 x upper limits of normal (ULN) OR measured or calculated creatinine clearance (per institutional standard) must be >= 45 ml/min (obtained =< 15 days prior to registration)
* Total bilirubin =<1.5 x ULN OR direct bilirubin =< ULN for patients with total bilirubin levels >1.5 x ULN (obtained =< 15 days prior to registration)
* Aspartate transaminase (AST) AND alanine transaminase (ALT) =< 2.5 x ULN (obtained =< 15 days prior to registration)
* Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) =< 1.5 x ULN OR if patient is receiving anticoagulant therapy then INR or aPTT is within target range of therapy (obtained =< 15 days prior to registration)
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only (POCBP) Note: If testing done for eligibility is > 72 hours prior to first dose, then pregnancy testing must be repeated, and result must be negative for patient to receive treatment.
* POCBP or able to father a child must be willing to use adequate contraception starting with first dose through 180 days after last dose
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study).
* Willing to provide tissue and blood samples for correlative research purposes

Exclusion Criteria:

* Any of the following because this study involves an investigational agent for which genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential or able to father a child who are unwilling to employ adequate contraception
* Signs or symptoms of life-threatening raised intracranial pressure: as determined by the treating neurosurgeon, including severe headache, nausea, decreasing level of consciousness, precluding 4-7-day delay in scheduling neurosurgery (i.e., immediate surgery is indicated, and patient cannot wait).
* Prior treatment

  * Received bevacizumab (AVASTIN) =< 4 months prior to registration

    * Note: Bevacizumab is allowed for symptom control during the adjuvant phase of the study
  * Received a live vaccine =< 30 days prior to registration.
  * Requirement for dexamethasone dose of > 2mg/day =< 2 days prior to registration
* Failure to recover from any adverse events related to any of the following therapies received prior to registration:

  * Major surgery =< 28 days prior to registration
  * Radiation therapy =< 14 days prior to registration
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Known history of human immunodeficiency virus (HIV) infection
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations (e.g., drug addiction) that would limit compliance with study requirements
* Receiving any other investigational agent
* Other active malignancy requiring systemic treatment =< 1 year prior to registration
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Active autoimmune disease that has required systemic treatment (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) =< 2 years prior to registration NOTE: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Concurrent known active Hepatitis B (i.e., known positive hepatitis B virus [HBV] surface antigen [HBsAg] reactive) AND known active Hepatitis C (i.e., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] detected by polymerase chain reaction [PCR])

  * Note: No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority
  * NOTE: Patients with known Hepatitis B OR Hepatitis C may be enrolled if they meet the following criteria:

    * Hepatitis B: Patients who are HBsAG positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization. Patients should remain on anti-viral therapy throughout the treatment phase of the trial and should follow local guidelines for HBV anti-viral therapy after completing study treatment
    * Hepatitis C: Patients with history of Hepatitis C infection are eligible if HCV viral load is undetectable at screening. Patients must have completed curative anti-viral therapy at least 4 weeks prior to registration
* Known history of active TB (Bacillus Tuberculosis)
* History of (non-infectious) pneumonitis or interstitial lung disease that required steroids, or current pneumonitis or interstitial lung disease
* Hypersensitivity to pembrolizumab or any of its excipients
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent within < 12 months prior to registration

  * NOTE: If such therapy was given ≥ 12 months prior to registration, patient is eligible
* History of allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-10-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | Up to 9 months
  9-month overall survival rate (OS9) rate is defined as the number of "successes" (patients who are alive at least 9 months after beginning study therapy) divided by the total evaluable patients. All patients who have signed a consent form, are eligible, and have begun treatment in Cycle 1 (first cycle of neo-adjuvant pembrolizumab + efineptakin alfa [NT-I7]) will be considered evaluable for the primary endpoint.

SECONDARY OUTCOMES:
Progression free survival time | From the date of starting study treatment to the date of disease progression or death resulting from any cause, whichever comes first, assessed up to 5 years
  Progression is defined according to Immunotherapy Response Assessment in Neuro-Oncology (iRANO) criteria. The median and 95% confidence intervals will be estimated using the Kaplan-Meier estimator.
Objective response rate (ORR) | Up to 5 years
  Objective response rate (ORR) is defined as the number of responses achieved during treatment with pembrolizumab + NT-I7 in combination with surgery divided by the total number of evaluable patients. A patient will be deemed to have a response if complete response (CR) or partial response (PR) is achieved. Only patients with measurable disease documented on the post-operative baseline scan (prior to initiation of Cycle 2) will be considered evaluable for ORR. Point estimates will be generated for response rate with corresponding 95% binomial confidence intervals (Duffy and Santner).
Changes in absolute lymphocyte counts (ALC) | From baseline up to 12 weeks
  Point estimates will be generated for the difference (at the magnitude of a fold-change) with corresponding 95% confidence intervals. All other changes in ALC over time will be exploratory and hypothesis generating. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Incidence of adverse events | Up to 5 years
  The number and severity of all adverse events will be tabulated and summarized in this patient population. Specifically, the overall percentages for Grade 3 or higher adverse events considered at least possibly related to treatment will also be calculated and reported. All other adverse event analysis will be exploratory and hypothesis generating. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Jian L. Campian, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials